CLINICAL TRIAL: NCT03336060
Title: Long-term Effects of ACL Reconstruction Surgery on Neurophysiologic Correlates of Movement Planning During Complex Jump Landing Tasks and the Role of Neuropsychological Performance Measures: An Explorative Cross-sectional Study
Brief Title: Neurophysiologic Correlates of Movement Planning During Complex Jump Landing Tasks and the Role of Cognitive Function
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Goethe University (Other)
Responsible Party: Principal Investigator, Prof. Dr. Dr. Winfried Banzer, Head of Department, Dpt. Sports Medicine, Goethe University
Other Study IDs: SpM2016-006
Record Dates: First submitted 2017-10-27; First posted 2017-11-08 (Actual); Last update posted 2018-03-15 (Actual); Status verified 2018-03

CONDITIONS: Anterior Cruciate Ligament Reconstruction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Control: Age matched healthy subjects. Inclusion criteria for healthy controls are: male (18 - 40 years, right-handed); sportive (preferably ball game sports, e.g. soccer); no acute injury or life-quality impairing diseases; no medication
  Interventions: Diagnostic Test: Cortical Correlates of Jump Landing Task
- Subjects with ACL reconstruction: Unilateral, primary anterior cruciate ligament tear and reconstruction (1 to 10 years ago); no serious concomitant injuries, e.g. "unhappy triad"); no kinesiophobia; symmetric single leg jump performance (>85 %); male (18 - 40 years, right-handed); sportive (preferably ball game sports, e.g. soccer); no acute injury or life-quality impairing diseases; no medication
  Interventions: Diagnostic Test: Cortical Correlates of Jump Landing Task

INTERVENTIONS:
Diagnostic Test: Cortical Correlates of Jump Landing Task — The study participants perform counter-movement jumps (CMJ, flight time approximately 500 ms) followed by single leg landings. While under an anticipated condition, the individuals receive the visual information (presented on a screen) on which leg/ foot (left, right) they are required to land before self-initiated CMJs, the individuals will receive this information under the non-anticipated condition only after take-off (approximately 400 ms before ground contact).

SUMMARY:
To examine the long-term effects of anterior cruciate ligament injuries and reconstructions (after successful rehabilitation) on cortical processes of motor planning during complex jump landing tasks and the relevance of cognitive performance measures for landing stability, respectively knee injury risk.

DETAILED DESCRIPTION:
Particularly, in the context of ball sports ruptures of the anterior cruciate ligament (ACL) are among the most frequent injuries. However, the ACL tear does not only result in a loss of mechanical stability in the knee joint: the tear of the ligament and the subsequent reconstructive surgery lead to a massive damage of so-called mechanoreceptors (proprioceptors). These small sensors provide the brain with precise information on the tension of the cruciate ligament and the position of the knee joint. Due to this feedback, it is possible for humans to adjust the activity of the stabilizing muscles to various situations in sports and daily life and to protect the knee from injuries. Thus, coordination deficits are common consequences after ACL-rupture and reconstruction due to the poorer sensory feedback.

New findings provide evidence that the injury-induced damage of the mechanoreceptors also causes persistent, neuronal reorganisations in the brain (injury induced neuroplasticity). These relate in particular to the motor cortex by which voluntary movements are controlled. According to the results of imaging (eg. functional magnetic resonance tomography; MRI) and electrophysiological studies (eg. Electroencephalography; EEG), these neurologic adaptation appear to persist far beyond the resumption of daily, sporting or competitive activities. Researchers suggest that these adaptations of the central nervous system might be the underlying cause of the frequently observed, persistent motor control and functional deficits (eg. muscle strength and muscle activation deficits), the relatively high re-injury, low return to sports rates and small proportions returning to their initial performance level after ACL tears and reconstruction. A pure restoration of the neuromuscular function without the elimination of the neuroplastic changes in the brain does therefore not appear sufficient.

In recent studies the effects of ACL trauma on brain activity have been investigated exclusively during unspecific, sport- and injury-unrelated tests (eg. simple flexion and extension movements and angular reproduction tasks of the knee). Often, injuries to the ACL occur under unpredictable conditions, especially in complex, dynamic movements such as changes of direction, jumps and landings. Here, the brain has to process information from the receptors of the ACL as quickly as possible to initiate an adequate motor response to protect the knee.

Against the background of the above described findings, this cross-sectional case-control study will firstly investigate the effects of completely healed ACL tears and reconstruction (side symmetry of neuromuscular performance measures above 85%) on movement planning related cortical activity (via Electroencephalography) measures during complex jump-landing tasks: The study participants perform counter-movement jumps (n=80; CMJ, flight time approximately 500 ms) followed by single leg landings. While under an anticipated condition (n=40), the individuals receive the visual information (presented on a screen) on which leg/ foot (left, right) they are required to land before self-initiated CMJs, the individuals will receive this information under the non-anticipated condition (n=40) only after take-off (approximately 400 ms before ground contact). The measurement of the landing stability is standardized by means of selected biomechanical parameters (capacitive force platform). Injury-relevant, cognitive characteristics (e.g., reaction, information processing speed and working memory) are detected by computer and paper-based clinical cognition tests.

The investigators hypothesize that the injury-related neurological adjustments in the motor cortex lead to a more intensive motor action planning before movement initiation (compensation of sensory deficits). The increased use of neuronal capacities for movement planning could subsequently lead to a slower or to unprecise motor responses to unforeseen/ non-anticipated events and subsequently cause greater landing instability, or increase the knee injury risk, respectively. It is also assumed that a lower cognitive information processing is associated with a more instable landing, or a higher risk of injury or higher injury incidence rate, respectively.

ELIGIBILITY:
Inclusion Criteria:

* male (18 - 40 years, right-handed)
* sportive (preferably ball game sports, e.g. soccer)

Only cases:

* unilateral, primary anterior cruciate ligament tear and reconstruction (1-10yrs ago)
* no serious concomitant injuries (e.g. "unhappy triad")
* no kinesiophobia
* symmetric single leg jump performance (>85 %)

Exclusion Criteria:

* acute injury or life-quality impairing diseases
* any medication

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Cases: Healthy male participants (18 - 40 lifeyears) with unilateral ACL reconstruction and succesfull rehabilitation Controls: Healthy male participants (18 - 40 lifeyears)
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-05-31 (Estimated); Study Completion 2018-06-30 (Estimated)

PRIMARY OUTCOMES:
Bereitschaftspotential - Movement planning associated cortical activity measures | Cross sectional design. Time Frame for Assessment of Movement planning associated cortical activity measures (Bereitschaftspotential, low beta-band power, frontal theta-band power) is 4 hours on one day
  Determined via Electroencephalography as amplitude in microvolt [μV] and latency in milliseconds [ms] before initiation of jump movement
Sensorimotor rhythm (SMR)/ low beta-band power - Movement planning associated cortical activity measures | Cross sectional design. Time Frame for Assessment of Movement planning associated cortical activity measures (Bereitschaftspotential, low beta-band power, frontal theta-band power) is 4 hours on one day
  Determined via Electroencephalography in microvolt^2 [μV²]
Frontal theta-band power - Movement planning associated cortical activity measures | Cross sectional design. Time Frame for Assessment of Movement planning associated cortical activity measures (Bereitschaftspotential, SMR/ low beta-band power, frontal theta-band power) is 4 hours on one day
  Determined via Electroencephalography in microvolt^2 [μV²]

SECONDARY OUTCOMES:
Peak ground reaction force - Biomechanical outcome measures of single leg jump-landings | Cross sectional design. Biomechanical outcome measures of single leg jump-landings are assessed simultaneously with primary outcome assessment (during same 4 hours on one day)
  Determined via capacitive force platform: Biomechanical outcome measure of single leg jump-landing (Newton [N])
Time to stabilisation - Biomechanical outcome measures of single leg jump-landings | Cross sectional design. Biomechanical outcome measures of single leg jump-landings are assessed simultaneously with primary outcome assessment (during same 4 hours on one day)
  Determined via capacitive force platform: Biomechanical outcome measure of single leg jump-landing (seconds [s])
Center of pressure sway - Biomechanical outcome measures of single leg jump-landings | Cross sectional design. Biomechanical outcome measures of single leg jump-landings are assessed simultaneously with primary outcome assessment (during same 4 hours on one day)
  Determined via capacitive force platform: Biomechanical outcome measure of single leg jump-landing (in millimeter [mm])^2 [μV²])
Visual perceptual ability - Lower cognitive function | Cross sectional design. Timeframe for Assessment is 5 minutes (during congnitive function assessment, separate day as primary outcome assessment)
  Determined via pen and paper tests: Trail Making Test A (Time for task completion in seconds [s])
Reaction time/ processing speed - Lower cognitive function | Cross sectional design. Timeframe for Assessment is 10 minutes (during congnitive function assessment, separate day as primary outcome assessment)
  Determined via computer-based neuropsychological test (mean of the log10 transformed reaction times for correct responses in milliseconds [ms])
Working memory - Higher cognitive function | Cross sectional design. Timeframe for Assessment is 10 minutes (during congnitive function assessment, separate day as primary outcome assessment)
  Determined via computer-based neuropsychological test (One card learning test: Speed of performance (mean of the log10 transformed reaction times for correct responses) and Accuracy of performance (arcsine transformation of the square root of the proportion of correct responses); Digit Span Task: Number of correct reproduced digits)
Cognitive flexibility - Higher cognitive function | Cross sectional design. Timeframe for Assessment is 5 minutes (during congnitive function assessment, separate day as primary outcome assessment)
  Determined via pen and paper test: Trail-Making-Test B vs. A (time for task completion in seconds [s])
Inhibitory control - Higher cognitive function | Cross sectional design. Timeframe for Assessment is 15 minutes (during congnitive function assessment, separate day as primary outcome assessment)
  Determined via computer-based neuropsychological test: Stop-Signal-Task (Stop signal reaction time in milliseconds [ms])
Interference control - Higher cognitive function | Cross sectional design. Timeframe for Assessment is 5 minutes (during congnitive function assessment, separate day as primary outcome assessment)
  Determined via pen and paper test: Stroop-Test (Time for task completion in seconds [s])
Kinesiophobia (subjective measure) - Potential confounder | Cross sectional design. Time Frame for Assessments is 5 minutes (same day as cognitive function assessment)
  Determined via questionnaire (Tampa scale)
Self-reported knee function (subjective measure) - Potential confounder | Cross sectional design. Time Frame for Assessments is 5 minutes (same day as cognitive function assessment)
  Determined via questionnaire (Lysholm knee score)
Physical activities (subjective measure) - Potential confounder | Cross sectional design. Time Frame for Assessments is 5 minutes (same day as cognitive function assessment)
  Determined via questionnaire (IPAQ)
Sport activities (current and past; subjective measure) - Potential confounder | Cross sectional design. Time Frame for Assessments is 5 minutes (same day as cognitive function assessment)
  Determined via questionnaire
Risk behaviour (subjective measure) - Potential confounder | Cross sectional design. Time Frame for Assessments is 5 minutes (same day as cognitive function assessment)
  Determined via questionnaire (DOSPERT scale)
Musculoskeletal injuries (current and past; subjective measure) - Potential confounder | Cross sectional design. Time Frame for Assessments is 5 minutes (same day as cognitive function assessment)
  Determined via questionnaire
Single and both legs jump performance (objective measure) - Potential confounder | Cross sectional design. Time Frame for Assessments is 5 minutes (same day as cognitive function assessment)
  Determined via motor testing (in centimeter [cm])
Single leg jump symmetry (objective measure) - Potential confounder | Cross sectional design. Time Frame for Assessments is 5 minutes (same day as cognitive function assessment)
  Determined via motor testing (in percent [%])
Static postural control (objective measure) - Potential confounder | Cross sectional design. Time Frame for Assessments is 5 minutes (same day as cognitive function assessment)
  Determined via motor testing (in millimeter [mm])
Visuomotor reaction time (objective measure) - Potential confounder | Cross sectional design. Time Frame for Assessments is 5 minutes (same day as cognitive function assessment)
  Determined via computer-based neuropsychological test (in milliseconds [ms])

CONTACTS AND LOCATIONS:
Overall Officials: Winfried Banzer, Prof, Principal Investigator — Head of Department; Goethe University Department of Sports Medicine
Locations (1):
- Goethe University Department of Sports Medicine, Frankfurt am Main, Hesse, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Giesche F, Engeroff T, Wilke J, Niederer D, Vogt L, Banzer W. Neurophysiological correlates of motor planning and movement initiation in ACL-reconstructed individuals: a case-control study. BMJ Open. 2018 Sep 19;8(9):e023048. doi: 10.1136/bmjopen-2018-023048. PMID 30232114